CLINICAL TRIAL: NCT05410535
Title: A Multi-center, Phase IV, Extension Study in PEGASUS-D Trial to Evaluate Efficacy of Ursodeoxycholic Acid (UDCA) for the Prevention of Gallstone Formation After Gastrectomy in Patients With Gastric Cancer
Brief Title: To Evaluate Efficacy of Ursodeoxycholic Acid (UDCA) for the Prevention of Gallstone Formation After Gasterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DW_UDCA005_P401
Record Dates: First submitted 2021-12-22; First posted 2022-06-08 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Dosage Forms; Prescriptions

STUDY DESIGN:
Intervention Model Description: patients who participated in PEGASUS-D clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients who received UDCA 600mg (Experimental): Patients who participated in PEGASUS-D clinical trial and received UDCA 600mg
  Interventions: Drug: Patients who continued UDCA 300mg medication; Other: Patients who discontinued UDCA 300mg prescription
- Patients who received UDCA 300mg (Experimental): Patients who participated in PEGASUS-D clinical trial and received UDCA 300mg
  Interventions: Drug: Patients who continued UDCA 300mg medication; Other: Patients who discontinued UDCA 300mg prescription
- Patients who received Placebo (Placebo Comparator): Patients who participated in PEGASUS-D clinical trial and received Placebo
  Interventions: Drug: Patients who continued UDCA 300mg medication; Other: Patients who discontinued UDCA 300mg prescription

INTERVENTIONS:
Drug: Patients who continued UDCA 300mg medication — patients who continued UDCA 300mg prescription for the prevention of gallstone after PEGASUS-d trial
Other: Patients who discontinued UDCA 300mg prescription — patients who discontinued UDCA 300mg prescription for the prevention of gallstone after PEGASUS-d trial

SUMMARY:
Of those patients who participated in PEGASUS-D FAS clinical trial, patient must sign the informed consent form in order to participate in this extension study.

The medical records of the patients will be reviewed throughout the study.

DETAILED DESCRIPTION:
Of those patients who participated in PEGASUS-D FAS clinical trial, patient must sign the informed consent form in order to participate in this extension study.

* Collection of retrospective cohort data

  1)The medical records from the subject's gastrectomy surgery date to Visit1 will be collected through a questionnaire and by reviewing the medical records of the patient.
* Collection of prospective cohort data

  1. Based on visit 1, if the subjects whose date of gastrectomy surgery date is more than 3 years(36 months) and less than 5 years(60 months), the subject should visit the institution at the time of 5 years(60 months, visit2) after gastrectomy surgery to evaluate data requested at visit2.
  2. The medical records will be accessed and collected from the subject's gastrectomy surgery date up to 5 years(60 months)

ELIGIBILITY:
Inclusion Criteria:

Among the PEGASUS-D Full Analysis Set (FAS) subjects, those who agree to participate in this clinical trial or those who can collect retrospective cohort data after waiving consent according to the consent waiver criteria

Exclusion Criteria:

A person who, at the discretion of the investigator, is deemed difficult to participate in this clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with gallstones formed | at 3 years
  The proportion of subjects with gallstones formed after gastrectomy.
Proportion of subjects with gallstones formed | at 5 years
  The proportion of subjects with gallstones formed after gastrectomy.
The incidence of symptomatic gallstones, acute cholecystitis, cholangitis, pancreatitis, liver abscess, and cholecystectomy. | at 3 years
  The incidence of symptomatic gallstones, acute cholecystitis, cholangitis, pancreatitis, liver abscess, and cholecystectomy.
The incidence of symptomatic gallstones, acute cholecystitis, cholangitis, pancreatitis, liver abscess, and cholecystectomy. | at 5 years
  The incidence of symptomatic gallstones, acute cholecystitis, cholangitis, pancreatitis, liver abscess, and cholecystectomy.
The duration of UDCA | up to 5 years
  The duration of UDCA
The dose of UDCA | up to 5 years
  The dose of UDCA
The recurrence rate of gastric cancer | up to 5 years
  The recurrence rate of gastric cancer
The survival rate of gastric cancer | up to 5 years
  The survival rate of gastric cancer

CONTACTS AND LOCATIONS:
Overall Officials: DoJoong Park, Principal Investigator — Seoul National University Hospital
Locations (1):
- DoJoong Park, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided